CLINICAL TRIAL: NCT06454344
Title: Associations of Adverse Childhood Experiences, Sleep Disruption, and Vascular Dysfunction in Young Adults: The Iowa ACEs and Sleep Cohort and Manipulating Sleep in Young Adults With ACEs Studies
Brief Title: The Iowa ACEs and Sleep Cohort and Manipulating Sleep in Young Adults With ACEs Studies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nathaniel Jenkins (Other)
Responsible Party: Sponsor-Investigator, Nathaniel Jenkins, Assistant Professor, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 202307139; 1R01HL167788-01A1 (NIH)
Record Dates: First submitted 2024-06-03; First posted 2024-06-12 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Adverse Childhood Experiences; Vascular Dilatation; Sleep; Sleep Disturbance; Psychosocial Stressor; Psychological Trauma; Endothelial Dysfunction; Inflammation; Oxidative Stress
MeSH Terms: conditions — Aneurysm; Parasomnias; Psychological Trauma; Inflammation | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy for Insomnia (CBT-i) (Experimental)
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-i)
- Waitlist Control (No Intervention)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-i) — CBT-I is a structured program with a robust empirical evidence supporting its efficacy for improving sleep quality and quantity. The cognitive component of CBT-I teaching individuals how to recognize and change the beliefs they hold about sleep that negatively impact sleep, such as negative thoughts and emotions. The behavioral component includes several strategies to help improve sleep, including: improved sleep hygiene, improving the sleep environment, relaxation training, stimulus control therapy (consistent wake/sleep times, using the bed only for sleep, etc), and sleep restriction. Sleep restriction consists of reducing the time spend in bed initially to increase sleep drive in subsequent nights. Once sleep has improved, the time in bed is gradually increased again.
  Arms: Cognitive Behavioral Therapy for Insomnia (CBT-i)

SUMMARY:
The overall purpose of this study is to understand the role of disrupted sleep in the association of exposure to early life adversity (adverse childhood experiences (ACEs)) with vascular endothelial (dys)function.

In Aim 1 (The Iowa ACEs and Sleep Cohort Study), the investigators will utilize a cross-sectional cohort design with a state-of-the-art translational approach. Participants will be recruited to objectively characterize the degree to which lower sleep quality and quantity contribute to ACEs-related endothelial dysfunction, inflammation, and oxidative stress in young adults using:

1. rigorous at home sleep monitoring using 7-nights of wrist actigraphy and 2 nights of home-based polysomnography to objectively measure sleep quality (sleep efficiency, wakefulness after sleep onset and sleep depth), and total sleep duration,
2. in vivo assessment of endothelial function via flow-mediated dilation testing, and
3. in vitro determination of endothelial cell inflammation and oxidative stress from biopsied endothelial cells. This study to achieve this Aim.

In Aim 2, approximately 70 eligible participants from Aim 1 (The Iowa ACEs and Sleep Cohort Study) will then be randomized to either a 6-week behavioral sleep intervention (cognitive behavioral therapy for insomnia) or a wait-list control to determine the mechanistic contribution of sleep disruption to vascular dysfunction in young adults with moderate-to-high exposure to adverse childhood experiences (ACEs). Following the intervention, participants will again complete:

1. rigorous at home sleep monitoring using 7-nights of wrist actigraphy and 2 nights of home-based polysomnography to objectively measure sleep quality (sleep efficiency, wakefulness after sleep onset and sleep depth), and total sleep duration,
2. in vivo assessment of endothelial function via flow-mediated dilation testing, and
3. in vitro determination of endothelial cell inflammation and oxidative stress from biopsied endothelial cells.

ELIGIBILITY:
AIM 1

Inclusion Criteria:

1. 18-29 years of age
2. SBP <129 and DBP <90 mmHg
3. Body Mass Index > 18.5 kg/m2 and <35 kg/m2
4. Willing to complete in-home sleep studies

Exclusion Criteria:

1. Currently undergoing treatment for a sleep disorder or diagnosed with restless leg syndrome, hypersomnia, parasomnia or narcolepsy, or obstructive sleep apnea
2. Currently performing overnight shift work
3. Lifetime history of any psychiatric disorder with psychotic features or bipolar disorder, currently undergoing treatment for substance-induced mood disorder
4. Endorsed suicidal ideation as indicated by a Moderate or High risk determination on the Columbia Suicide Risk Protocol
5. Diagnosed neurological disorder or illness affecting the central nervous system
6. Diagnosed acute or chronic autoimmune disease or chronic inflammatory condition
7. Current or previous cancer diagnosis
8. History of moderate or severe traumatic brain injury
9. Current or previous history of CBT-I treatment or sleep restriction or cognitive restructuring therapy for sleep
10. History of cardiometabolic disease (e.g., ischemic heart disease, coronary artery disease, stroke, chronic kidney disease, diabetes mellitus), pulmonary disease, or renal disease
11. Current or recent (within past month) use of anti-hypertensive (including clonidine), lipid lowering, glucose- controlling, or prescription anti-inflammatory medications
12. Current or recent (within past month) opiates, benzodiazepine or benzodiazepine receptor agonists, or trazodone
13. Recent changes to or unstable treatment (changes within last 6 mo.) with prescription medications
14. Currently smoking or using nicotine
15. Current use of hormone therapy
16. Current heavy alcohol use, as defined as binge drinking on 5 or more days in the last month, or consuming more than 7 (women) or 14 (men) drinks per week in the last month (per NIAAA definition)
17. Current or recent (within the last 6 mo.) illicit drug use disorder as indicated by a score of 3 or greater on the Drug Abuse Screening Test (DAST-10)
18. Current or recent (within 6 mo.) pregnancy OR current or recent breastfeeding (within 3 mo.) OR children under the age of 2 years old in the home
19. Currently completing greater than 300 minutes of moderate intensity, or greater than 150 minutes of vigorous intensity physical activity, or an equal combination per week
20. Unstable housing

AIM 2

Inclusion Criteria:

1. 18-29 years of age
2. SBP <129 and DBP <90 mmHg
3. Body Mass Index > 18.5 kg/m2 and <35 kg/m2
4. Willing to complete in-home sleep studies
5. >= 3 Adverse Childhood Experiences
6. PSQI Global Score >5
7. Sleep Efficiency Score <90%

Exclusion Criteria:

1. Currently undergoing treatment for a sleep disorder or diagnosed with restless leg syndrome, hypersomnia, parasomnia or narcolepsy, or obstructive sleep apnea
2. Currently performing overnight shift work
3. Lifetime history of any psychiatric disorder with psychotic features or bipolar disorder, currently undergoing treatment for substance-induced mood disorder
4. Endorsed suicidal ideation as indicated by a Moderate or High risk determination on the Columbia Suicide Risk Protocol
5. Diagnosed neurological disorder or illness affecting the central nervous system
6. Diagnosed acute or chronic autoimmune disease or chronic inflammatory condition
7. Current or previous cancer diagnosis
8. History of moderate or severe traumatic brain injury
9. Current or previous history of CBT-I treatment or sleep restriction or cognitive restructuring therapy for sleep
10. History of cardiometabolic disease (e.g., ischemic heart disease, coronary artery disease, stroke, chronic kidney disease, diabetes mellitus), pulmonary disease, or renal disease
11. Current or recent (within past month) use of anti-hypertensive (including clonidine), lipid lowering, glucose- controlling, or prescription anti-inflammatory medications
12. Current or recent (within past month) opiates, benzodiazepine or benzodiazepine receptor agonists, or trazodone
13. Recent changes to or unstable treatment (changes within last 6 mo.) with prescription medications
14. Currently smoking or using nicotine
15. Current use of hormone therapy
16. Current heavy alcohol use, as defined as binge drinking on 5 or more days in the last month, or consuming more than 7 (women) or 14 (men) drinks per week in the last month (per NIAAA definition)
17. Current or recent (within the last 6 mo.) illicit drug use disorder as indicated by a score of 3 or greater on the Drug Abuse Screening Test (DAST-10)
18. Current or recent (within 6 mo.) pregnancy OR current or recent breastfeeding (within 3 mo.) OR children under the age of 2 years old in the home
19. Currently completing greater than 300 minutes of moderate intensity, or greater than 150 minutes of vigorous intensity physical activity, or an equal combination per week
20. Unstable housing
21. Likely Obstructive Sleep Apnea, as indicated by an apnea-hypopnea index (AHI) >= 15 events/hour or persistent hypoxemia, as indicated by an arterial oxygen saturation <= 88% for >5 minutes per night.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Vascular Endothelial Function | Week 0 (Pre-Intervention) and Week 7 (Post-Intervention)
  The brachial artery flow-mediated dilation (FMD) technique, a non-invasive bioassay of endothelium-dependent vasodilatory function, will be used as the primary determinant of in-vivo vascular endothelial function.

SECONDARY OUTCOMES:
Endothelial NFκB p65 expression. | Week 0 (Pre-Intervention) and Week 7 (Post-Intervention)
  Vascular endothelial cells will be biopsied and stained for inflammatory marker NFκB p65.
Endothelial TNF-α expression. | Week 0 (Pre-Intervention) and Week 7 (Post-Intervention)
  Vascular endothelial cells will be biopsied and stained for inflammatory marker TNF-α.
Endothelial MCP-1 expression. | Week 0 (Pre-Intervention) and Week 7 (Post-Intervention)
  Vascular endothelial cells will be biopsied and stained for inflammatory marker MCP-1.
Endothelial NADPH-oxidase p47phox expression. | Week 0 (Pre-Intervention) and Week 7 (Post-Intervention)
  Vascular endothelial cells will be biopsied and stained for NADPH-oxidase p47phox, a marker of oxidative stress.
Endothelial nitrotyrosine expression. | Week 0 (Pre-Intervention) and Week 7 (Post-Intervention)
  Vascular endothelial cells will be biopsied and stained for nitrotyrosine, a marker of oxidative stress.
Circulating CRP | Week 0 (Pre-Intervention) and Week 7 (Post-Intervention)
  Blood samples will be collected and analyzed for inflammatory marker CRP in plasma.
Circulating TNF-α | Week 0 (Pre-Intervention) and Week 7 (Post-Intervention)
  Blood samples will be collected and analyzed for inflammatory marker TNF-α in serum.
Circulating MCP-1 | Week 0 (Pre-Intervention) and Week 7 (Post-Intervention)
  Blood samples will be collected and analyzed for inflammatory marker MCP-1 in serum.
Circulating IL1-RA | Week 0 (Pre-Intervention) and Week 7 (Post-Intervention)
  Blood samples will be collected and analyzed for inflammatory marker IL1-RA in plasma.
Circulating oxidized low density lipoprotein | Week 0 (Pre-Intervention) and Week 7 (Post-Intervention)
  Blood samples will be collected and analyzed for oxidative stress marker oxidized low density lipoprotein in serum.
Circulating 8-iso prostaglandin F2α | Week 0 (Pre-Intervention) and Week 7 (Post-Intervention)
  Blood samples will be collected and analyzed for oxidative stress marker 8-iso prostaglandin F2α in serum.
Anti-oxidant (Superoxide Dismutase) Activity in Peripheral Blood Mononuclear Cells | Week 0 (Pre-Intervention) and Week 7 (Post-Intervention)
  Peripheral blood mononuclear cells will be isolated from whole blood pre and post intervention and superoxide dismutase activity will be quantified using calorimetric assay.
Anti-oxidant (Glutathione Reductase) Activity in Peripheral Blood Mononuclear Cells | Week 0 (Pre-Intervention) and Week 7 (Post-Intervention)
  Peripheral blood mononuclear cells will be isolated from whole blood pre and post intervention and glutathione reductase activity will be quantified using calorimetric assay.
Anti-oxidant (Catalase) Activity in Peripheral Blood Mononuclear Cells | Week 0 (Pre-Intervention) and Week 7 (Post-Intervention)
  Peripheral blood mononuclear cells will be isolated from whole blood pre and post intervention and catalase activity will be quantified using calorimetric assay.
Perceived Stress | Week 0 (Pre-Intervention) and Week 7 (Post-Intervention)
  The investigators will measure perceived stress using the "Perceived Stress Scale" (PSS-10). This will be considered one of the mediators alongside sleep in the investigators' models, as the addition of other potential mediators can improve power and provide a more accurate estimate of the original (sleep) mediator by controlling for shared effects among mediators. The PSS-10 has a minimum score of "0" and a maximum score of "40" with higher scores indicating worse outcomes.
Distress | Week 0 (Pre-Intervention) and Week 7 (Post-Intervention)
  The investigators will measure distress using the "Kessler Psychological Distress Scale" (K-10). This will be considered one of the mediators alongside sleep in the investigators' models, as the addition of other potential mediators can improve power and provide a more accurate estimate of the original (sleep) mediator by controlling for shared effects among mediators. The K-10 has a minimum score of "10" and a maximum score of "50" with higher scores indicating worse outcomes.

OTHER OUTCOMES:
Sleep Quality | Week 0 (Pre-Intervention) and Week 7 (Post-Intervention)
  The investigators will objectively quantify sleep quality as actigraphy measured as sleep efficiency (PRIMARY independent variable) and wakefulness after sleep onset and PSG measured sleep depth as indicated by the relative time spent in slow wave sleep. The investigators will also assess sleep efficiency and wakefulness after sleep onset using sleep diaries. These parameters are considered the independent variable in this study, with the primary identified independent variable identified as sleep efficiency. Collection of these data will be used to a) confirm changes and b) examine whether changes in the variables do in fact mediate changes in vascular function.
Sleep Duration | Week 0 (Pre-Intervention) and Week 7 (Post-Intervention)
  The investigators will objectively quantify total sleep duration using actigraphy and via sleep diary.
Anxiety and Depression | Week 0 (Pre-Intervention) and Week 7 (Post-Intervention)
  Anxiety and depression symptoms will be assessed using the "Inventory of Depression and Anxiety Symptoms-II" (IDAS-II), which is a reliable, well-validated assessment of mood and anxiety disorder symptoms. Using this scale, anxiety and depression ill be well-measured, and the investigators will assess their role as confounders/mediators in analyses. Each scale is individually assessed, meaning that the minimum score for mood symptoms, specifically, ranges from 3-20, and the maximum score ranges from 15-100 for this scale. With regards to anxiety disorder symptoms, the minimum score ranges from 3-8, and the maximum score ranges from 15-40. Higher scores on scales indicate worse outcomes.
Trauma | Week 0 (Pre-Intervention) and Week 7 (Post-Intervention)
  Trauma symptoms will be assessed using the "PTSD Checklist for DSM-5" (PCL-5) with Life Events checklist. Using this scale, trauma symptoms will be well-measured, and the investigators will assess their role as confounders/mediators in analyses. The minimum value for this scale is "0" and the maximum value for this scale is "80". Higher scores on this scale indicate a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Jenkins, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Integrative Laboratory of Applied Physiology and Lifestyle Medicine, Iowa City, Iowa, United States

DOCUMENTS (2):
  • Statistical Analysis Plan (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/44/NCT06454344/SAP_000.pdf
  • Informed Consent Form (2024-05-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT06454344/ICF_001.pdf